CLINICAL TRIAL: NCT01450930
Title: Pharmacokinetics of Hydrocortisone After Subcutaneous Administration Compared With Intramuscular Injection in Chronic Adrenal Insufficiency
Brief Title: Pharmacokinetics of Hydrocortisone After Subcutaneous Administration in Chronic Adrenal Insufficiency
Acronym: PHYSCA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bruno Allolio (Other)
Responsible Party: Sponsor-Investigator, Bruno Allolio, MD, Professor of Medicine, head of the Dept. of Endocrinology and Diabetology, University of Wuerzburg, University of Wuerzburg
Organization: University of Wuerzburg (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PHYSCA-1; 2011-002687-25 (EudraCT Number)
Record Dates: First submitted 2011-09-29; First posted 2011-10-13 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Primary Adrenal Insufficiency
Keywords: Adrenal insufficiency; Addison's disease
MeSH Terms: conditions — Addison Disease; Adrenal Insufficiency | interventions — Hydrocortisone; Solvents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrocortisone subcutaneously first (Active Comparator): Hydrocortisone subcutaneously first
  Interventions: Drug: Hydrocortisone subcutaneously first
- Hydrocortisone intramuscular first (Active Comparator): Hydrocortisone intramuscular first
  Interventions: Drug: Hydrocortisone intramuscular first

INTERVENTIONS:
Drug: Hydrocortisone intramuscular first — Hydrocortisone intramuscular first
  Other Names: 100 mg hydrocortisone (Pfizer®) in 2 ml solvent
  Arms: Hydrocortisone intramuscular first
Drug: Hydrocortisone subcutaneously first — Hydrocortisone subcutaneously first
  Other Names: 100 mg hydrocortisone (Pfizer®) in 2 ml solvent
  Arms: Hydrocortisone subcutaneously first

SUMMARY:
Patients with chronic adrenal insufficiency need to adapt their hydrocortisone replacement dose in conditions of physical or psychological stress to prevent life threatening adrenal crisis. In cases of more severe impairment or unsecure gastrointestinal absorption (e.g. gastroenteritis, severe infectious disease), parenteral administration of the hydrocortisone dose is crucial. The study is conducted to offer patients the possibility to perform hydrocortisone self administration in emergency situations in a way of administration which is easy to perform and accepted by the patient. Therefore, pharmacokinetics and safety of subcutaneous hydrocortisone administration will be studied and compared to intramuscular administration.

ELIGIBILITY:
Inclusion Criteria:

* Primary adrenal insufficiency under standard glucocorticoid replacement therapy due to autoimmune adrenalitis or bilateral adrenalectomy (disease duration at least 12 months),
* age ≥ 18 years,
* Patient´s written informed consent,
* Ability to comply with the protocol procedures

Exclusion criteria

* Diabetes mellitus,
* Infectious disease with fever at time of investigation,
* Known intolerance to the study drug or constituents oft he study drug,
* Oral contraception,
* Known pregnancy or breast feeding,
* Renal failure (creatinine > 2.5 ULN)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence Study | 4 hours
  pharmakokinetic data (Cmax, time to Cmax, area under the curve of serum/salivary cortisol levels)

SECONDARY OUTCOMES:
safety | 3 days
  number of adverse events after subcutaneous administration of hydrocortisone

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Hahner, MD, Principal Investigator — University Hospital Wuerzburg, Germany
Locations (1):
- Dept of Medicine I, Endocrinology and Diabetology, University Hospital Wuerzburg, Würzburg, Germany

REFERENCES:
- [Derived] Hahner S, Burger-Stritt S, Allolio B. Subcutaneous hydrocortisone administration for emergency use in adrenal insufficiency. Eur J Endocrinol. 2013 Jun 29;169(2):147-54. doi: 10.1530/EJE-12-1057. Print 2013 Aug. PMID 23672956